CLINICAL TRIAL: NCT04679012
Title: Phase II Study of Polatuzumab Vedotin in Combination With Chemotherapy in Subjects With Richter's Transformation
Brief Title: Polatuzumab Vedotin in Combination With Chemotherapy in Subjects With Richter's Transformation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-08022533
Record Dates: First submitted 2020-12-16; First posted 2020-12-22 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Richter Syndrome; Chronic Lymphocytic Leukemia
Keywords: Polatuzumab vedotin; CLL; Richter's Transformation
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — polatuzumab vedotin; Rituximab; Etoposide; etoposide phosphate; Prednisone; Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Polatuzumab vedotin plus R-EPCH (Experimental): Polatuzumab vedotin will be given in conjunction with 6 cycles of R-EPCH (rituximab, etoposide, prednisone, cyclophosphamide, hydroxydaunorubicin). The dosing schedule and regimen for R-EPCH will follow established protocols. Polatuzumab vedotin will be administered on Day 1 of each 21-day cycle.
  Interventions: Drug: Polatuzumab Vedotin; Drug: Rituximab; Drug: Etoposide; Drug: Prednisone; Drug: Cyclophosphamide; Drug: Hydroxydaunomycin

INTERVENTIONS:
Drug: Polatuzumab Vedotin — Polatuzumab vedotin will be administered as an IV infusion at 1.8mg/kg on Day 1 of each cycle, every 21 days.
  Other Names: Polivy
Drug: Rituximab — Rituximab will be obtained from commercial supply, and will be given for a total of 6 cycles for all patients. The drug will be given by IV route.
  Other Names: Rituxan; chimeric anti-CD20 monoclonal antibody
Drug: Etoposide — Etoposide will be obtained from commercial supply, and will be given for a total of 6 cycles for all patients. The drug will be given by IV route.
  Other Names: VP-16; VePesid; etopophos; toposar
Drug: Prednisone — Prednisone will be obtained from commercial supply, and will be given for a total of 6 cycles for all patients. Prednisone will be given orally.
  Other Names: Deltasone; Orasone; Paracort; Cortan
Drug: Cyclophosphamide — Cyclophosphamide will be obtained from commercial supply, and will be given for a total of 6 cycles for all patients. The drug will be given by IV route.
  Other Names: cytoxan
Drug: Hydroxydaunomycin — Hydroxydaunomycin will be obtained from commercial supply, and will be given for a total of 6 cycles for all patients. The drug will be given by IV route.
  Other Names: Doxorubicin Hydrochloride; Hydroxydoxorubicin Hydrochloride

SUMMARY:
This study evaluates the effectiveness and safety of Polatuzumab vedotin plus infusional chemoimmunotherapy containing rituximab, etoposide, prednisone, cyclophosphamide and hydroxydaunorubicin. This is a single arm study. Enrolled patients will receive up to six cycles (21-day cycles) of therapy. While on study, subjects will be monitored weekly until end of treatment, then followed for 52 weeks or until disease progression or discontinuation due to toxicity or death. After completion of the 52-week follow-up/End of study visit, Subjects will be followed for an additional 104 week period, with an assessment occurring every 12 weeks to evaluate survival outcomes and next line of treatments only.

DETAILED DESCRIPTION:
This is an open label, single arm, phase II investigator initiated clinical trial, evaluating efficacy and safety of Polatuzumab vedotin added to a modified infusional dose adjusted R-EPOCH like regimen, given on an inpatient basis, every 21 days, in subjects with Richter's Transformation.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have confirmed diagnosis of CLL or small lymphocytic lymphoma (SLL) based upon 2018 International Workshop on CLL (IwCLL) criteria, with biopsy proven Richter's Transformation to a DLBCL subtype.
* Subject must be ≥18 years of age.
* Subject must be able to sign informed consent
* Ability and willingness to comply with the study protocol procedures
* Life expectancy of at least 24 weeks
* Subject must have an Eastern Cooperative Oncology Group performance status of ≤2.
* Subject must have measurable disease with atleast on LN>- 1.5cm in longest diameter
* Subject must have adequate bone marrow function and meet the below thresholds prior to treatment.

  * Absolute neutrophil count of ≥1000 cell/uL
  * Hemoglobin ≥ 7 g/dL
  * Platelet count ≥ 30,000 cells/uL- Subjects may receive growth factor or transfusion support no less than 7 days prior to enrollment or C1 D1.
* Subject must have adequate organ function and meet the thresholds below:

  * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN). Subjects with Gilbert's disease will be granted exception to this rule.
  * Creatinine clearance >30 ml/min/1.73m2 as calculated by the MDRD equation.
  * Ejection fraction ≥ 50% measured by transthoracic echocardiogram or MUGA scan
* For women of childbearing potential: agreement to remain abstinent or use of contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 12 months after the last dose of study drug.

  * A woman is considered to be of childbearing potential if she is post-menarcheal, has not reached a postmenopausal state (i.e. ≥ 12 months of amenorrhea with no identified cause other than menopause) and has not undergone surgical sterilization (removal of ovaries and or uterus)

    * Acceptable forms of contraception are bilateral tubal ligation, male sterilization, or copper intrauterine devices.
  * For women considered to have childbearing potential a negative serum pregnancy test within 7 days prior to study enrollment and dosing is required.
* For men, agreement to remain abstinent, or to use a condom plus an additional contraceptive method during the treatment period and for at least 5 months after the last dose of study drug.

  * Men must agree not to donate sperm during that period of time. Male patients interested in preservation of fertility should be advised to sperm bank prior to enrollment and treatment initiation.

Exclusion Criteria:

* Diagnosis of Richter's Transformation not of DLBCL subtype (including but not limited to Hodgkin lymphoma, PLL)
* Prior therapy targeting Richter's transformation.
* Any subject that initiates a targeted agent such as BTKi, venetoclax, or PI3K prior to enrollment (Continuation of a targeted CLL directed therapy such as a BTKi, venetoclax, or PI3K will be permitted as a bridge through screening but add on therapies or change in therapy will be exclusionary. These continuation therapies will be permitted up 72 hours prior to study initiation. Bridging therapy with steroid up to equivalent of 40mg of Dexamethasone daily will be allowed prior to study treatment and can be continued up to 24 hours prior to study treatment)
* Subject has undergone an allogeneic stem cell transplant for CLL within 6 months of study entry.
* Subject has an active or presumed secondary malignancy at time of enrollment. A subject will be eligible if a previous malignancy was treated with curative intent and there is no evidence of disease recurrence for the past 3 years. Non-melanomatous and cervical squamous cell cancers are an exception and if excised will be allowed to enroll regardless of timing of excision.
* Subject is known to be positive for HIV.
* Active hepatitis C or hepatitis B defined by positive PCRs for viral DNA/RNA. Subjects with a positive Hep B core antibody and negative PCR, are allowed to enroll (prophylaxis is strongly encouraged and monthly monitoring of Hep B PCR is mandatory).
* Subject has baseline ≥ Grade 2 or greater peripheral neuropathy.
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Clinical evidence or known central nervous system involvement with transformed large cells
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results
* Significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, congestive heart failure, myocardial infarction within the previous 6 months, unstable arrhythmias, or unstable angina)
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection requiring treatment with intravenous antibiotics or hospitalization within 4 weeks before Cycle 1 day 1.
* Major surgery within 4 weeks before the start of Cycle 1 day 1. Superficial lymph node biopsies or laprascopic lymph node biopsies are exclusionary to this rule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Complete metabolic remission/complete remission (CMR/CR) rate of subjects at end of treatment (EOT) | 19 weeks
  Percentage of subjects who achieve CMR/CR on study.

SECONDARY OUTCOMES:
Safety of polatuzumab vedotin plus infusional chemoimmunotherapy (CIT) containing rituximab, etoposide, prednisone, cyclophosphamide and hydroxydaunorubicin in patients with newly diagnosed Richter's Transformation. | 1.5 years
  Percentage of subjects who experience 1 or more adverse events.
Overall response rate (ORR) | 3 years
  Rate of subjects who achieve a partial or complete response.
Progression free survival (PFS) | 3 years
  Measured from time of first study drug administration to objective or symptomatic progression or death.
Overall survival (OS) | 3 years
  Measured from time of first study drug administration to death from any cause.
Allogeneic transplantation rate in eligible patients | 3 years
  Percentage of eligible patients able to get allogeneic stem cell transplant.

CONTACTS AND LOCATIONS:
Overall Officials: John Allan, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - Mount Sinai- Icahn School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Ohio state University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: WCM Joint Clinical Trials Office — http://jcto.weill.cornell.edu/